CLINICAL TRIAL: NCT04460586
Title: Pharmacokinetics of Omadacycline in Patients With Cystic Fibrosis
Brief Title: Pharmacokinetics of Omadacycline in Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Paul Beringer (Other)
Collaborators: Paratek Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor-Investigator, Paul Beringer, Professor of Clinical Pharmacy, University of Southern California
Organization: University of Southern California (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS-20-00513
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — omadacycline

STUDY DESIGN:
Intervention Model Description: A single group of patients with CF will receive a single dose of omadacycline 100mg IV followed by a 1-week washout and receipt of 300 mg PO.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omadacycline IV followed by PO (Experimental): Omadacycline 100mg IV, Omadacycline 300 mg tablet
  Interventions: Drug: Omadacycline Injection [Nuzyra]; Drug: Omadacycline Oral Tablet [Nuzyra]

INTERVENTIONS:
Drug: Omadacycline Injection [Nuzyra] — Participants will receive single dose of omadacycline 100mg IV followed by a 1-week washout and receipt of single dose omadacycline 300 mg PO.
Drug: Omadacycline Oral Tablet [Nuzyra] — Participants will receive single dose of omadacycline 100mg IV followed by a 1-week washout and receipt of single dose omadacycline 300 mg PO.

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics of intravenous and oral omadacycline in patients with cystic fibrosis.

DETAILED DESCRIPTION:
Omadacycline exhibits excellent activity against bacteria including methicillin-resistant Staphylococcus aureus (MRSA), Burkholderia cepacia, and Nontuberculous mycobacteria (NTM) that are a potential source of lung infection in CF patients. As omadacycline demonstrates antimicrobial activity against a number of pathogens in CF, the investigators hope to learn the optimal dose of omadacycline necessary to treat lung infections in patients with CF in the future. The study hypothesis is that omadacycline will exhibit good oral bioavailability in patients with CF.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF based on positive sweat chloride or known CF mutation
* Age >=18 years

Exclusion Criteria:

* Presence of an ongoing acute pulmonary exacerbation defined based on clinical signs & symptoms and an acute decline in relative FEV1 of 10% or greater.
* Pregnancy or breastfeeding
* Serious past allergy to a tetracycline antibiotic
* No alcohol, nicotine, or caffeine-containing products during the study period
* Hemoglobin < 8 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cmax | 3 Days
  To assess the maximum concentration of omadacycline after single dose of oral and intravenous administration.
Tmax | 3 days
  To assess the time to maximum concentration of omadacycline after single dose of oral and intravenous administration.
AUC | 3 days
  To assess the area under the plasma concentration time curve of omadacycline after single dose of oral and intravenous administration.
Absolute Bioavailability | 6 days
  To determine the absolute bioavailability of omadacycline following single dose of IV and PO administration.

CONTACTS AND LOCATIONS:
Overall Officials: Adupa P Rao, M.D., Study Director — Keck Medicine of USC
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Sanders M, Hong E, Chung PS, Rao AP, Beringer P. Pharmacokinetics of Omadacycline in Adults with Cystic Fibrosis. Clin Pharmacokinet. 2024 Dec;63(12):1701-1709. doi: 10.1007/s40262-024-01440-w. Epub 2024 Nov 24. PMID 39581957